CLINICAL TRIAL: NCT00151892
Title: A Phase III, Randomized Multi-centre, Double-blind, Parallel Group, Active Comparator Study to Compare the Efficacy and Safety of SPD476 (Mesalazine)2.4g/Day Once Daily With Asacol 1.6g/Day Twice Daily in the Maintenance of Remission in Patients With Ulcerative Colitis
Brief Title: Efficacy and Safety of SPD476 in Maintaining Remission in Patients With Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD476-304; 2004-004184-29 (EudraCT Number)
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Results first posted 2010-09-21 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- SPD476 (Experimental): Mesalazine
  Interventions: Drug: SPD476
- Asacol (Active Comparator)
  Interventions: Drug: Asacol

INTERVENTIONS:
Drug: SPD476 — 2.4 g/day Once Daily (QD)
  Other Names: Lialda; mesalazine; mesalamine; MMX mesalamine
  Arms: SPD476
Drug: Asacol — 1.6g/day administered 800 mg Twice Daily (BID)
  Other Names: mesalamine
  Arms: Asacol

SUMMARY:
Ulcerative colitis is a disease of the large bowel (colon) and rectum in which the lining of the bowel becomes red and swollen. Over time, patients with this disease may experience acute episodes of diarrhea, rectal bleeding and abdominal pain followed by periods of time without disease symptoms. 5-ASA drugs are a standard treatment for ulcerative colitis. Mesalazine is an experimental drug designed to gradually release 5-ASA into the areas of large bowel associated with ulcerative colitis. This study will test the safety and efficacy of mesalazine in keeping ulcerative colitis in remission.

ELIGIBILITY:
Inclusion Criteria:

* previous diagnosis of ulcerative colitis confirmed by histology that has been considered to be in remission for => 30 days
* female subjects must be post-menopausal, surgically or biologically sterile, or with a negative urine pregnancy test at screening and on adequate contraception

Exclusion Criteria:

* proctitis
* previous resective colonic surgery
* Crohn's disease
* hypersensitivity to salicylates
* moderate/severe renal impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 829 (Actual)
Dates: Start 2005-04-08 (Actual); Primary Completion 2009-09-07 (Actual); Study Completion 2009-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (141):
- United States (15):
  - Birmingham Gastroenterology Associates, Birmingham, Alabama
  - Connecticut Gastroenterology Institute, Bristol, Connecticut
  - Washington Gastroenterology, Washington D.C., District of Columbia
  - Southern Clinical Research Consultants, Hollywood, Florida
  - Boorland-Groover Clinic, Jacksonville, Florida
  - United Medical Research, New Smyrna Beach, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Midwest Clinical Research Center, Moline, Illinois
  - Gastrointestinal Clinic of Quad Cities, Davenport, Iowa
  - Drug Research Services, Inc., Metairie, Louisiana
  - Mayo Clinic, Rochester, Minnesota
  - Center for Digestive and Liver Diseases, Inc, Mexico, Missouri
  - New York Center for Clinical Research, Lake Success, New York
  - ClinSearch, Chattanooga, Tennessee
  - S D Khan, Houston, Texas
- Argentina (3):
  - Hospital Italiano de Buenos Aires, Capital Federal, Buenos Aires
  - Centro Integral De Gastroenterologia, Ciudad de Buenos Aires
  - Hospital Italiano de Mendoza, FINAMED SA, Mendoza
- Australia (6):
  - Bankstown-Lidcombe Hospital, Bankstown, New South Wales
  - Concord Hospital, Concord, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Eastern Health Hospital, Box Hill, Victoria
  - St Vincent's Hospital, Fitzroy, Victoria
  - Fremantle Hospital, Fremantle, Western Australia
- Belgium (3):
  - Imelda General Hospital, Bonheiden
  - Ziekenhuis Oost Limburg, Genk
  - Heilig Hart ziekenhuis vzw Roeselare-Menen, Roeselare
- Brazil (6):
  - Unigastro, Castelo
  - Hospital de Clinicas, Porto Alegre
  - Universidade Federal do Rio de Janeiro, Rio de Janeiro
  - Universidade Federal da Bahia - Hospital, Salvador
  - Hospital Sao Paulo, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo
- Canada (5):
  - University of Calgary, Calgary, Alberta
  - Toronto Digestive Disease Associates, Inc., Toronto, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Hópital Hótel-Dieu de Quebec, Québec, Quebec
  - GI Research, Edmonton
- Chile (4):
  - Hospital del Salvador, Santiago
  - Clinica Las Condes, Santiago
  - Hospital Clinico P.UC, Santiago
  - Hospital San Juan de Dios, Santiago
- Czechia (9):
  - Fakultni Nemocnice Plzen, Pilsen
  - NZZ Online 24 s.r.o, Prague
  - Remedis s.r.o, Prague
  - Thomavers Hospital, Prague
  - Klinicke Centrum ISCARE I.V.F, Prague
  - Nemocnice Jablonec nad Nisou p.o, Prague
  - Oblastni Nemocnice Pribram, Příbram
  - Nemocnice Tabor A.S., Tábor
  - Masarykova Nemocnice, Ústí nad Labem
- Denmark (3):
  - Bispebjerg Hospital, Copenhagen NV
  - Hvidovre Hospital, Hvidovre
  - Koge University Hospital, Køge
- France (3):
  - CHU de Grenoble, Grenoble
  - Hospital De L'Archet, Nice
  - Hospital Haut Leveque, Pessac
- Germany (3):
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - Universitat des Saarlandes, Homburg
  - Gastroenterologische Praxis Prof. Hackelsberger, Wiesbaden
- Hungary (5):
  - Peterfy Sandor utcai, Budapest
  - Semmelweis Egyetem, Budapest
  - Debreceni Egyetem OEC - III, Debrecen
  - Markhot Ferenc Korhaz-Rendelointeze II. Belgyogyaszat - Gasztroenterologia, Eger
  - Pandy Kalman County Hospital, Gyula
- India (9):
  - Amrita Institute of Medical Sciences, Kochi, Kerala
  - Lifeline Multispeciality Hospital, Chennai
  - Asian Institute of Gastreoenterology, Hyderabaad
  - S.R. Kalla Memorial Gastro & General Hospital, Jaipur
  - Sanjay Gandhi Post Graduate Institute of Medical Sciences, Lucknow
  - Dayanand Medical College and Hospital, Ludhiana
  - Jaslok Hospital and Research Centre, Mumbai
  - All India Institute of Medical Sciences, New Delhi
  - Sree Gokulam Medical Centre & Research Foundation, Trivandrum
- Mexico (6):
  - Unidad Medica de Endoscopia y Cirugia (UNIMEDEC), La Paz, Baja California Sur
  - Hospital San Javier, Guadalajara
  - Central de Especialidades Medicas (FIDEPAZ), La Paz
  - Mexican Institute of Clinical Research, Mexico City
  - Instituto Nacional de Ciencias médicas y Nutrición Salvador Zubirán, Mexico City
  - Hospital Angeles Torreón, Torreón
- Netherlands (2):
  - Orbis Medical Centre, Sittard
  - Isala Clinics, Zwolle
- New Zealand (4):
  - Shakespeare Specialist Group, Auckland
  - Waikato DHB Hospital, Hamilton
  - Tauranga Hospital BOP Medical, Tauranga
  - Wellington Hospital, Wellington
- Peru (4):
  - Hospital Nacional Edgardo Rebagliati Martins, Lima
  - Hospital Nacional Guillermo Alemnara Irigoyen, Lima
  - Clinica Anglo America, Lima
  - Clinica El Golf, Lima
- Poland (5):
  - Klinika Gastroenterologi, Bialystok
  - Klinika Gastroenterologii, Lodz
  - Klinika Gastroenterologii, Szczecin
  - Miejska Przychodnia Specjalistyczna, Torun
  - Katedra i Klinika Gastroenterologii, Warsaw
- Portugal (3):
  - Hospital Sao Marcos, Braga
  - Hospital Egas Moniz, Lisbon
  - Hospital Geral Santo Antonio, Porto
- Romania (6):
  - Colentina Clinical Hospital, Bucharest
  - Prf. Dr D. Gerota Emergency Hospital, Bucharest
  - Octavian Fodor Clinical Emergency Hospital, Cluj-Napoca
  - County Emergency Hospital, Constanța
  - Institute of Gastronenterology & Hepatology, Iași
  - Clinical County Emergency Hospital, Târgu Mureş
- Russia (5):
  - City Hospital #24, Moscow
  - City Hospital #51, Moscow
  - Scientific Centre of Coloproctology, Moscow
  - City Hospital #122, Saint Petersburg
  - Russian Academy of Sciences, Saint Petersburg
- Singapore (3):
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
  - Changi General Hospital, Singapore
- South Africa (8):
  - Louis Leipoldt Medical Centre, Bellville, Western Cape
  - New Groote Schuur Hospital, Observatory, Western Cape
  - Kingsbury Hospital, Cape Town
  - St Augustine's Hospital, Durban
  - Parklands Medical Centre, Durban
  - Milpark Hospital, Johannesburg
  - Greenacres Hospital, Port Elizabeth
  - 2H Arun Place, Somerset West
- South Korea (6):
  - Hallyam University, Sacred Heart Hospital, Anyang-si
  - Seoul National University Hospital, Seoul
  - Samsung Medical Centre, Seoul
  - The Catholic University of Korea Kangnam St Mary's Hospital, Seoul
  - Asan Medical Center, Seoul
  - Yonsei University, College of Medicine, Seoul
- Spain (4):
  - Hospital Universitario Germans Trias I Pujol, Badalona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital de Sagunto, Valencia
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Sophiahemmet, Stockholm
  - Karolinska University Hospital, Stockholm
- Taiwan (3):
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (5):
  - St. Mark's Hospital, Harrow, Middlesex
  - Addenbrookes Hospital Department of Gastroenterology, Cambridge
  - Imperial College School of Medicine, London
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Royal Hallamshire Hospital, Sheffield

REFERENCES:
- See also: FDA-approved label — http://www.lialda.com/Professional/pdf/pi.pdf
- See also: FDA recall information — http://www.fda.gov/opacom/7alerts.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SPD476 | Asacol
Started | 416 | 413
Completed | 340 | 330
Not Completed | 76 | 83
Not completed — Lack of Efficacy | 50 | 57
Not completed — Patient request | 10 | 7
Not completed — Lost to Follow-up | 5 | 10
Not completed — Adverse Event | 6 | 3
Not completed — Protocol Violation | 3 | 3
Not completed — Non-compliance | 0 | 1
Not completed — Pregnancy | 0 | 1
Not completed — Did not return for a visit | 1 | 0
Not completed — Used prohibited corticosteroids | 1 | 0
Not completed — Lack of study medication at center | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- SPD476: 2.4 g/day QD
- Asacol: 1.6g/day administered 800 mg BID
- Total: Total of all reporting groups
Arm/Group | SPD476 | Asacol | Total
Number analyzed (Participants) | 415 | 411 | 826
Age, Continuous [Mean (Standard Deviation); unit: years] — Baseline characteristics were calculated from the Safety Population (n = 826) defined as all randomized subjects who received at least 1 dose of investigational product.
  years | 45.0 (14.05) | 45.2 (13.44) | 45.1 (13.74)
Age, Customized [Count of Participants; unit: Participants] — Baseline characteristics were calculated from the Safety Population (n = 826) defined as all randomized subjects who received at least 1 dose of investigational product.
  Participants
    <18 years | 0 | 0 | 0
    18 to 64 years | 380 | 377 | 757
    >=65 years | 35 | 34 | 69
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline characteristics were calculated from the Safety Population (n = 826) defined as all randomized subjects who received at least 1 dose of investigational product.
  Participants
    Female | 203 | 197 | 400
    Male | 212 | 214 | 426
Region of Enrollment [Count of Participants; unit: Participants] — Baseline characteristics were calculated from the Safety Population (n = 826) defined as all randomized subjects who received at least 1 dose of investigational product.
  Participants
    United States | 24 | 22 | 46
    Taiwan | 1 | 0 | 1
    Spain | 3 | 4 | 7
    Chile | 4 | 4 | 8
    Russian Federation | 51 | 49 | 100
    India | 81 | 83 | 164
    France | 2 | 3 | 5
    Denmark | 6 | 5 | 11
    Australia | 4 | 3 | 7
    Peru | 7 | 7 | 14
    South Africa | 18 | 17 | 35
    Netherlands | 1 | 0 | 1
    Korea, Republic of | 17 | 14 | 31
    United Kingdom | 7 | 7 | 14
    Hungary | 25 | 25 | 50
    Czech Republic | 50 | 54 | 104
    Mexico | 7 | 10 | 17
    Canada | 15 | 14 | 29
    Argentina | 4 | 2 | 6
    Brazil | 25 | 28 | 53
    Belgium | 11 | 11 | 22
    Poland | 29 | 31 | 60
    Singapore | 3 | 4 | 7
    Romania | 11 | 10 | 21
    Germany | 2 | 1 | 3
    New Zealand | 4 | 2 | 6
    Sweden | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Endoscopic Remission of Ulcerative Colitis (UC) at 6 Months
Description: Endoscopic remission is defined as an endoscopy score of less than or equal to 1. Endoscopy score (mucosal appearance) ranges from 0-3 (0 = normal [intact vascular pattern; no friability or granulation], 1 = mild [erythema; decreased vascular pattern; minimal granularity], 2 = moderate [marked erythema; granularity; friability; absent vascular pattern; bleeding with minimal trauma; no ulcerations], 3 = severe [ulceration; spontaneous bleeding].
Time Frame: 6 Months
Population: Per Protocol Population (PP) defined as all subjects who either completed the study or withdrew for reasons related to efficacy or AEs and who were deemed to be protocol-compliant.
Measure: Number; unit: percent of participants
Arm/Group | SPD476 | Asacol
Number analyzed (Participants) | 343 | 336
percent of participants | 83.7 | 81.5
Statistical Analysis 1: Comparison: SPD476 vs Asacol; The null hypothesis to be tested is that the true difference in proportions is less than or equal to -10%; Test type: Non-Inferiority or Equivalence — A 2-sided 95% confidence interval (CI) for the difference in the percentages of subjects in remission at 6 months of the two treatment groups will be computed. Non-inferiority of SPD476 to Asacol will be concluded if the lower limit of the 95% CI lies above the non-inferiority margin of -10%; Difference in proportions = 0.02, 95% CI [-0.04 to 0.08]

2. Secondary Outcome: Withdrawal Due to Relapse of UC
Description: Relapse is defined as withdrawal from the study due to lack of efficacy.
Time Frame: Over 6 Months
Population: PP
Measure: Number; unit: percent of participants
Arm/Group | SPD476 | Asacol
Number analyzed (Participants) | 343 | 336
percent of participants | 12.8 | 14.6

3. Secondary Outcome: Endoscopic Remission of UC With No or Mild Symptoms at 6 Months
Description: Endoscopic remission with no or mild symptoms is defined as an endoscopy score of less than or equal to 1 and a combined symptom score (stool frequency plus rectal bleeding) of less than or equal to 1. Endoscopy score (mucosal appearance) ranges from 0-3 (0 = normal, 1 = mild , 2 = moderate, 3 = severe). Rectal bleeding is assessed on a scale from 0-3 (0 = no rectal bleeding, 1 = streaks of blood, 2 = obvious blood, 3 = mostly blood). Stool frequency is assessed on a scale of 0-2 (0 = 0-1 more than normal per day, 1 = 2-3 more than normal per day, 2 = 4 or more than normal per day).
Time Frame: 6 Months
Population: PP
Measure: Number; unit: percent of participants
Arm/Group | SPD476 | Asacol
Number analyzed (Participants) | 343 | 336
percent of participants | 79.0 | 75.6

4. Secondary Outcome: Change From Baseline in Modified Ulcerative Colitis Disease Activity Index (UCDAI) Score at 6 Months
Description: The modified UCDAI score is the sum of the scores of 4 parameters (stool frequency, rectal bleeding, endoscopy score, and physician global assessment), each scoring between 0 and 3, making 12 the worst score.
Time Frame: Baseline and 6 months
Population: PP
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SPD476 | Asacol
Number analyzed (Participants) | 290 | 281
Units on a scale | 0.061 (1.1516) | 0.059 (1.2394)

5. Secondary Outcome: Short Inflammatory Bowel Disease Questionnaire (SIBDQ) Total Score
Description: Quality of life (QoL) was assessed using the SIBDQ. SIBDQ total score is calculated from the sum of 10 questions. Each question is scored on a scale from 1 (poor QoL) to 7 (good QoL) with total scores ranging from 10 to 70. Higher scores indicate better QoL.
Time Frame: 6 Months
Population: Intent to treat (ITT) population defined as all randomized subjects who received at least 1 dose of investigational product. Analysis includes patients who completed an SIBDQ questionnaire at 6 months.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SPD476 | Asacol
Number analyzed (Participants) | 155 | 155
Units on a scale | 59.523 (8.7582) | 59.664 (7.7440)

ADVERSE EVENTS:
Description: Safety population defined as all randomized subjects who received at least 1 dose of investigational medication.
Arm/Group | SPD476 | Asacol
Serious Adverse Events (participants affected / at risk) | 6/415 | 3/411
Other Adverse Events (participants affected / at risk) | 0/415 | 0/411
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SPD476 (N=415) | Asacol (N=411)
Colitis (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 1
Appendicitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Fallopian tube perforation (Injury, poisoning and procedural complications) | 0 | 1
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Radiculitis brachial (Nervous system disorders) | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.